CLINICAL TRIAL: NCT04402658
Title: The Effect of Inhaled Salbutamol on Sprint Performance During and After Submaximal Endurance Exercise in Non-asthmatic Athletes
Brief Title: Can Anti-asthmatic Medication Improve Sprint Performance in Healthy Endurance Athletes?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Problem with acquiring study medication and lack of resources.
Sponsor: Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Julie Stang, Principal Investigator, Norwegian School of Sport Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NorwegianSSS2020
Record Dates: First submitted 2020-04-29; First posted 2020-05-27 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Sports Drug Abuse
Keywords: Anaerobic performance; Athletes; Doping; Asthma; Endurance sports
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: The present study has a double-blinded and randomized cross-over design with participants visiting the laboratory on three separate occasions. The purpose of the first visit is to familiarize the participant with the equipment and the exercise performance protocol as well as to assess physiologic exercise data that will be used to determine the power output of the endurance exercise protocol on visits two and three. For a given participant, trials on day two and three will be conducted in randomized order, on the same time of day, and separated by more than 72 hours to ensure complete wash-out of salbutamol, and less than three weeks. The randomization will be performed using a computer random number generator.
Masking Description: Both participants and key study personnel will be blinded for the intervention as an external person will provide the participant with sequentially numbered drug containers of identical appearance, for salbutamol and placebo, respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physical performance test (Experimental): After performing measurements of lung function by spirometry, participants will inhale either salbutamol or placebo. After 15 minutes of rest, a second spirometry will be performed before the participants warm-up by 10 minutes cycling. The exercise protocol will consist of 60 minutes of cycling at 70% of maximal oxygen consumption (VO2max) on the cycle ergometer followed by an all-out sprint. Several times during the exercise test, 30-second Wingate tests will be conducted. Participants will be blinded to feedback such as power (W), distance covered, and heart rate. Strong verbal encouragement will be given to each participant for them to perform their best. Measurements of lung function (spirometry), heart rate, arterial oxygen saturation and Borg ratings of perceived exercising will be recorded throughout the trials, as well as capillary blood sampled for analysis of [La-] and [Glucose].
  Interventions: Drug: Inhaled salbutamol

INTERVENTIONS:
Drug: Inhaled salbutamol — Participants will inhale 800 μg salbutamol (or placebo) using a standard metered dose inhaler used for asthma treatment, and a standard spacer device will be used to allow optimal delivery of the drug to the lung. The inhaler delivers 100 μg of salbutamol with each actuation (i.e., 8 puffs/actuations gives 800 μg) with inhalation time being approximately ~2 min (10 breaths) and the manufacturer's user instructions will be followed. Although complete uptake of salbutamol cannot be concluded as any salbutamol left in the spacer, mouth or remaining in the lung will be not measured. This dose of Salbutamol is chosen because it is the highest dose permitted by the World Anti Doping Agency (WADA).

SUMMARY:
The prevalence of asthma among athletes is higher than in the normal population and endurance athletes are especially at increased risk. The gold standard for asthma treatment is inhaled glucocorticoids with inhaled beta2 agonists before exercise and as a symptom relief. However, the use of beta2 agonists in sports is debated because of potential performance-enhancing effects and its use is regulated by the World Anti-Doping Agency (WADA).

The potential performance-enhancing effect of beta2 agonists on endurance performance and sprint performance has each been investigated in several studies as it has been suspected that non-asthmatic athletes use beta2 agonists for the purpose of improving performance. In conclusion, beta2 agonists do not improve endurance athletic performance in the doses and methods of use permitted by WADA. When it comes to anaerobic performance, the evidence is currently non-conclusive as studies report conflicting effects. It is therefore conceivable that beta2 agonists can improve the ability to sprint and increase power output during short periods of high energy expenditure during an endurance competition. By testing such anaerobic skills during endurance work in athletes, this study will provide valuable knowledge about whether this drug may affect sports performance and will be of interest to WADA and anyone else interested in fair play in sports.

The purpose of the project is to investigate whether the use of a WADA approved dose of salbutamol (albuterol/Ventoline) has a performance-enhancing effect on sprint performance during and after endurance work on an ergometer bike. Well-trained cyclists who do not have asthma will perform two identical cycling protocols on two different days. The study is designed as a double-blind cross-over study with placebo. Participants will perform multiple 30-second sprints during a standard submaximal effort to investigate the effect of salbutamol on the maximum and average power of these sprints.

DETAILED DESCRIPTION:
Theoretical background:

The use of beta2-agonists in sports is restricted due to possible performance enhancing effects. The World Anti-Doping Agency's (WADA) prohibited list from January the 1st 2020 prohibits all use of beta2-agonists except inhaled salbutamol (maximum 1600 micrograms over 24 hours in divided doses not to exceed 800 micrograms over 12 hours starting from any dose), inhaled formoterol (maximum delivered dose of 54 micrograms over 24 hours) and inhaled salmeterol (maximum 200 micrograms over 24 hours).

Asthmatic athletes have consistently outperformed non-asthmatic athletes during the Olympic Games, and the use of inhaled beta2-agonists by athletes is surrounded by controversy, which have been highlighted in recent beta2-agonist anti-doping investigations involving world-class athletes. In 2020, Riiser et al. completed two systematic reviews with meta-analysis targeting the effect from beta2-agonists on aerobic (accepted in BSJM March 2020) and anaerobic (currently in review) performance. No effect was detected on aerobic performance, however an effect on anaerobic performance was reported. However, these meta-analyses separate the effects in either aerobic or anaerobic performance, while many sports requires both a high aerobic and anaerobic performance to succeed. For example, the development of endurance sports - such as cycling and cross-country skiing - has gone in a direction where anaerobic abilities are gaining importance, such as during sprints at the final stage of a race, closing gaps and during break away.

If beta2-agonists might improve performance in endurance sports through its effect on anaerobic performance, studies that better simulate this aspect of an endurance competitions is warranted. To the best of the present researcher's knowledge only three studies have investigated this aspect and they yielded conflicting results. In 1988, Bedi et al. found that competitive cyclists sprinted longer (196 sec vs 159 sec) after 60 min of cycling with a single inhalation of salbutamol pre-ride as compared to placebo. Furthermore, higher fatigue levels were reported during the final sprints after inhaling salbutamol, that may indicate a better ability to perform all-out anaerobic effort. However, Altarawneh et al. (2016) found no ergogenic effect of 1000 ug inhaled salbutamol on either continuous high-intensity (90 s at 130 % V̇O2max) performance or multiple sprint performance (3 sets of 5x4 s sprint with 20 s break between sprints and 4.5 min serial break) in recreationally active men. Fitness level has been suggested to confound the effect of beta2- agonists on physical performance, and to the best of our knowledge no study has investigated the effect of a WADA approved dose of inhaled salbutamol on measures of repeated bouts of anaerobic performance measured during prolonged submaximal exercise in well trained athletes. Therefore, because of the potential ergogenic effect of inhaled beta2-agonists on anaerobic performance combined with the potential reduced VO2 during submaximal work reported by Bedi et al. (1988), the combination of anaerobic performance and prolonged sub-maximal endurance exercise should be further investigated.

Materials and methods:

Participants eligible to the study will be recruited from local cycle and triathlon clubs, and sport high schools in the Oslo-area. The participants must be free from chest infection for at least 4 weeks prior to assessment; and are not to be taking any medication and have no other health or medical contradictions to them taking part in the study as confirm by information provided on a physical activity readiness questionnaire.

Participants will visit the laboratory on three separate occasions. Participants will be asked to prepare for each testing session in a similar manner and to refrain from caffeine and alcohol consumption and heavy exercise for 24 hours before the experiment.

Experimental procedures:

On the first visit to the laboratory, height and weight will be measured, and participants will fill out a physical activity readiness questionnaire before the test. Then the participants will complete an incremental step exercises test on a bicycle ergometer (Lode, Groningen, Netherlands) to establish the relationship between workload (W) and VO2. After a warmup phase, the workload will then increase by 25 watts every 5th minute with a pedal frequency of 90 revolutions per minute (rpm). During the last 3 min of each bout, VO2 (Oxycon Pro, Jaeger GmbH, Hoechberg, Germany) and heart rate (HR) (Polar, Kempele, Finland) will be measured. A capillary blood sample will be taken from a fingertip and analysed for blood lactate concentration [La-] (Biosen C-line, EKF diagnostic GmbH, Magdeburg, Germany) and glucose concentration [Glu] (HemoCue Glucose 201+, Ängholm, Sweden) after each 5 minutes bout of cycling. The test will be terminated when the participants reach a [la-] level of ≥1.5 mmolˑL-1 above baseline [La-]. Linear regression analysis from the incremental step exercise test will be used to determine the workload corresponding to 70% of VO2max for use on the same bicycle ergometer in the subsequent experimental trials. Participants will then immediately perform an incremental exercise test to determine VO2max. This test will start at the work rate (W) in the second last 5-min bout for each participant and the work rate will then be increased by 25 W each min, until exhaustion, defined as an inability to maintain pedal cadence above 60 rpm. After 20 minutes of rest, participants will perform 30-second Wingate tests for familiarisation purposes.

To exclude any participant with existing lung disease or asthma, the forced expiratory volume in 1 s (FEV1) and forced vital capacity (FVC) will be measured by spirometry using maximum expiratory flow volume loops (Oxycon Pro, Jaeger GmbH, Hoechberg, Germany) according to European standard before and 0, 3, 5 and 10 minutes after the VO2max test. In addition, on day 2 or 3 spirometry will be measured before and 15 minutes after inhalation of salbutamol of which can identify subjects with a bronchoconstriction (with a cut off at Δ FEV1 of ≥12% and 200 ml).

On day 2 and 3, identical protocols will be performed in randomized order as described elsewhere.

Questionnaires On day 1, the subjects will fill out a questionnaire regarding the type, duration, and intensity of training; exercise-related allergic and infectious symptoms; social habits (smoking); drug and food supplements intake and antidoping regulations (15). After each trial (day 2 and 3), participants will answer questions regarding respiratory symptoms, common side effects, sensations of dyspnoea and muscle fatigue, and if they can guess which intervention they received (salbutamol or placebo).

Statistical analyses Sample size is determined for the primary outcome "mean power" from the Wingate tests, as described by Dell, Holleran & Ramakrishnan (18). Effect size is based on the study by Collomp et al. (19) who reported a difference in mean power of 51 W after salbutamol (mean 585 +/- 27 W) vs placebo (534 +/- 35 W). Sample size calculations using an online a priori power calculator (https://clincalc.com/stats/samplesize.aspx) revealed that seven subjects in each group are necessary to obtain a power of 0.8 with a significance level of 0.05, and. With the risk of dropouts and to ensure a high statistical power with a lower salbutamol dose than in the study by Collomp et al., 20 participants will be included.

Two-way analyses of variance (ANOVA) for repeated measures will be used to evaluate the statistical significance of the variables measured. A Tukey post hoc test will be used to detect differences over time. A significance level (α) of 0.05 will be used.

Ethical considerations The study will be performed in accordance with the Declaration of Helsinki. Before recruiting participants, the Regional Ethical Committee should evaluate and approve the study. Written informed consent to take part will be obtained from participating athletes. Except for possible discomfort with tachycardia or shakiness, participants will not experience any expected side-effects.

Potential risks and benefits The investigators will include healthy, non-asthmatic participants that will be pre-screened for asthma by medical history, use of medication and lung function measured pre and post heavy exercise. The benefits of participation are that the participants will acquire measurements of their VO2max and blood lactate concentration during submaximal and maximal work which will be beneficial information for the athletes in terms of exercise planning. The participants may experience known side effects of inhaled salbutamol which include tremor, tachycardia, dry mouth, headache and muscle cramps (17). Adverse events (AE) will be reported to the primary investigator and the standard routines of the institution will be followed. This includes any event that is a result of a use error or intentional misuse (from ISO/FDIS 14155): any untoward medical occurrence, unintended disease or injury or any untoward clinical signs (including an abnormal laboratory finding) in participants, or other persons, related to the procedures involved (any procedure in the project plan).

Project responsibility and key roles The project will be carried out at the Norwegian School of Sport Sciences in Oslo, which will be the institution with the academic responsibility. Master students Martine Gøransson and Sandra Viksjø will perform the tests, under supervision by PhD Julie Stang, PhD Olav Vikmoen and PhD student Ove H Sollie. Prof. Thomas Halvorsen (MD) is medical responsible for the project. Professor Trine Stensrud and PhD Elisabeth Edvardsen are associate researchers in the project.

Data management Procedures for data management will be implemented according to the data processing routines at the Norwegian School of Sport Sciences and conducted according to standards of GCP. During the course of the study, the key investigators will have access to the study material, which will be secured by a data professional officer (DPO). Data will be de-identified and stored in a secured database. A Subject Identification List, with cross reference between the subject's identification number in the study and the subject's personal data, will be kept looked away with the study documentation. Only the key researchers will have access to this code book with the link between participant ID and data. Database cleaning and issuing data queries will be traceable and transparent with logs. Retention period for data storage is 5 years. Participating investigators will be responsible for data collection, data processing and report writing.

ELIGIBILITY:
Inclusion Criteria:

* well trained cyclists and triathletes (VO2max in mLˑkg-1ˑmin-1 ≥ 65 male/55 female) who are actively engaged in endurance cycling training at least 4 times per week.

Exclusion Criteria:

* a doctor diagnosed asthma and/or the use of anti-asthmatic medications the last 12 months prior to participation.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Anaerobic performance | Differences between experimental trial and placebo trial at 15 minutes
  Measures as mean power (Watts) from the 30-second Wingate tests carried out on an ergometer cycle.
Anaerobic performance | Differences between experimental trial and placebo trial at 30 minutes
  Measures as mean power (Watts) from the 30-second Wingate tests carried out on an ergometer cycle.
Sprint performance | Differences between experimental trial and placebo trial at 60 minutes
  Mean power (Watts) during an all-out sprint on an ergometer cycle.

SECONDARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) | Change from baseline FEV1 at 15 minutes
  Measurements of lung function by spirometry
Forced expiratory volume in 1 second (FEV1) | Change from baseline FEV1 at 30 minutes
  Measurements of lung function by spirometry
Forced expiratory volume in 1 second (FEV1) | Difference from placebo trial at 30 minutes
  Measurements of lung function by spirometry
Heart rate (btp) | Change from baseline heart rate at 15 minutes
  Heart rate measured by a Polar Chest-strap
Heart rate (btp) | Change from baseline heart rate at 30 minutes
  Heart rate measured by a Polar Chest-strap
Heart rate (btp) | Difference from placebo trial at 30 minutes
  Heart rate measured by a Polar Chest-strap

CONTACTS AND LOCATIONS:
Overall Officials: Julie S Stang, PhD, Principal Investigator — Norwegian School of Sport Sciences

IPD SHARING:
Plan to Share IPD: No